CLINICAL TRIAL: NCT06846658
Title: Exploring the Olfactory Mucosa, Blood and Urine for the Identification of Early Biomarkers of Parkinson's Disease, Atypical Parkinsonisms and Neurocognitive Disorders Due to Lewy Body Disease
Acronym: EXTRAORDINARY
Status: Recruiting | Type: Observational
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Other Study IDs: GR 2021 12372019
Record Dates: First submitted 2025-02-11; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease; MSA - Multiple System Atrophy; Lewy Body Dementia (LBD); Neurodegenerative Disease; Healthy Subjects (HS)
Keywords: Parkinson's disease (PD); multiple system atrophy (MSA); dementia with Lewy bodies (DLB); misfolded alpha-synuclein; new biomarkers; peripheral tissues; Real-Time Quaking-Induced Conversion (RT-QuIC); single-molecule array (Simoa); circulating neurofilament light chain (NfL); Nanoparticle Tracking Analysis (NTA); blood-derived extracellular vesicles (EVs); multi-omics analyses; transmission electron microscopy (TEM) and protein-NMR; protein misfolding; early diagnosis
MeSH Terms: conditions — Parkinson Disease; Shy-Drager Syndrome; Lewy Body Disease; Neurodegenerative Diseases; Multiple System Atrophy; Familial cylindromatosis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Clinical diagnosis of Parkinson's disease (PD), multiple system atrophy (MSA) and dementia with Lewy bodies (DLB) is challenging, especially in the early stages. Each disease is associated with distinct conformers of misfolded alpha-synuclein (maS) which form typical protein aggregates in the brain and represent key disease biomarkers. Thus, detection and characterization of intracerebral maS aggregates allow a definite diagnosis. The recent development of ultrasensitive assays enabled the detection of maS and other potential new biomarkers in peripheral tissues, although with several limitations. Here, the investigators propose to combine the expertise of leading and young researchers in the field of neurology, structural and molecular biology, biophysics and machine learning to perform ultrasensitive and multi-omics analyses of olfactory mucosa (OM), blood and urine of PD, MSA and DLB patients for detecting and characterizing key peripheral biomarkers allowing accurate disease recognition.

DETAILED DESCRIPTION:
OM, blood and urine likely contain key specific biomarkers of PD, MSA and DLB detectable with specialized ultrasensitive techniques, perhaps in the early disease stages. Therefore, by combining for the first time the RT-QuIC, Simoa SR-X, ELISA and NTA analyses of OM, blood and urine and by exploiting TEM and solution/solid-state NMR analyses, the investigators will attempt at identifying specific fingerprints of alpha-synucleinopathies usefult to stratify living patients. Supported by statistical analyses and customized machine learning algorithms that will combine clinical (including the analysis of olfactory functions) and experimental data, the investigators project could significantly impact the clinical diagnosis of alpha-synucleinopathies.

The investigators project will combine innovative and ultrasensitive diagnostic approaches to evaluate whether OM, blood and urine might serve as non-invasive and easy-to-get samples for biomarkers detection, allowing recognition and stratification of alpha-synucleinopathies. Multidisciplinary collaboration between researchers with specific and complementary skills is required to achieve the goals of the project and to have an impact on future scientific use, clinical applications and wellbeing of patients suffering from these diseases. The investigators project will combine cutting-edge technologies to improve the power of multidimensional biomarker patterns for the clinical diagnosis of PD, MSA and DLB by using easily and periodically collectible tissues. In particular, the investigators will determine unique insights into several key aspects of alpha-synucleinopathies by assessing whether: (1) the OM, blood and urine of PD, MSA and DLB patients contain peripheral maS exploitable to improve the patiens clinical diagnosis/recognition; (2) the peripheral distribution of maS in OM, blood and urine differs between diseases or even among tissues collected from the same patient; (3) the biochemical, morphological and structural features of the RT-QuIC generated aggregates enable discrimination of these diseases; (4) the levels of some key proteins (e.g. NfL, alpha-synuclein, synapsin-3) or structures (e.g. EVs), known to be altered in the blood, are also modified in the OM or urine and allow disease recognition, especially when analyzed in combination with the other ultrasensitive assays; (5) the olfactory impairment can be exploited as indicator of evolving alpha-synucleinopathy and whether it correlates with maS accumulation in OM. The investigators research is transformative and rapidly translatable into clinical practice. The possibility to accurately identify PD, MSA and DLB will bring important advancements in patient selection for emerging pharmacological treatments and clinical trials (better care for people). In addition, the possibility to periodically collect OM, blood and urine samples could consent to monitor disease progression and to evaluate the therapeutic effects in patients under pharmacological treatments. The Investigators findings could also contribute to further investigating whether PD, MSA and DLB are caused by distinct conformers of maS and verify if these latter possess differential tropism for peripheral tissues, eventually unveiling different molecular pathways involved in their pathogenesis. Finally, the investigators approach could have a major impact on counseling and prevention strategies for patients in the prodromal stages of alpha-synucleinopathies, representing a key goal on the path to disease-modifying and neuroprotective therapies before full-blown phenotypes have manifested.

ELIGIBILITY:
Inclusion Criteria:

* PD (Postuma et al., 2015), MSA (Palma et al., 2018), DLB (McKeith et al., 2017), OND including acquired and hereditary ataxic syndrome with known etiology, progressive supranuclear palsy, corticobasal degeneration, and motor neuron disease.

Exclusion Criteria:

* na

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: PD (n=20), MSA (n=20), DLB (n=20), OND (n=10, including acquired and hereditary ataxic syndrome with known etiology, progressive supranuclear palsy, corticobasal degeneration, and motor neuron disease) and HS (n=10).
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Identify a predictive model for the diagnosis of PD, MSA and DLB | 3 years
  To identify a predictive model for the diagnosis of PD, MSA and DLB based on the integration of:
  * Demographic and clinical: sex, age, comorbidities, disease duration and severity, current medications, cognitive status, the presence of bradykinesia, rigidity, tremors, orthostatic hypotension, autonomic failure, parkinsonism, visual hallucinations, cerebellar syndrome, dementia, rapid eye movement sleep behavior disorder;
  * Instrumental data: MRI, dopamine-transporter single-photon emission computerized tomography (DAT-SPECT), iodine-131-meta-iodobenzylguanidine (MIBG), fluorodeoxyglucose positron emission tomography (FDG-PET);
  * Results obtained from the biochemical, structural and RT-QuIC analyses of olfactory mucosa, blood and urine samples (gathered in detailed in the secondary outcomes measures paragraph).

SECONDARY OUTCOMES:
Analysis of olfactory functions. | 12 months
  To evaluate whether PD, DLB and MSA are characterized by different olfactory dysfunctions and if this can be exploited to discriminate the pathologies. Subjects will undergo olfactory evaluation by UPSIT test and divided in Normosmic, Hyposmic and Anosmic.
Evaluation of RT-QuIC accuracy in detecting maS in OM, blood- and urine-derived EVs | 21 months
  To study the distribution of maS in different peripheral tissues (urine, blood and olfactory mucosa) collected from the same patient with a clinical diagnosis of PD, MSA and DLB, by RT-QuIC.
Ultrasensitive detection and measurement of known or potential new biomarkers in OM, blood and urine of enrolled patients by Simoa SR-X. | 18 months
  To analyze if the levels of 181-p-tau (pg/mL), 231-p-tau (pg/mL) and neurofilament light chains (NfL, pg/mL) are altered in the biological samples analysed (urine, blood and OM) compared to subjects with non-neurodegenerative pathology (HS) and if these values differ in such a way as to discriminate the pathologies (PD, MSA and DLB). The assessment of these components will be pursued using Simoa SX-R.
Ultrasensitive detection and measurement of known or potential new biomarkers in OM, blood and urine of enrolled patients by ELISA. | 18 months
  To analyze if the levels of alpha-synuclein (pg/mL) and synapsin-III (pg/mL) are altered in the biological samples analysed (urine, blood and OM) compared to subjects with non-neurodegenerative pathology (HS) and if these values differ in such a way as to discriminate the pathologies (PD, MSA and DLB). These key proteins will be evaluated by ELISA.
NTA Nano-Sight NS300 analysis of concentration and size of EVs circulating in blood and urine. | 24 months
  To investigate whether the concentration (particles/mL and size distribution (nm)) of circulating EVs and the size features of rec-aS aggregates differ among PD, MSA, DLB patients, the other samples (b-EVs, u-EVs and rec-aS aggregates) will undergo NTA analysis.
Biochemical, morphological and structural characterization of selected RT-QuIC end products by Western blot and dot blot solution NMR and solid-state NMR analysis | 21 months
  To study if the RT-QuIC reaction products acquire biochemical (Western blot, Dot blot, densitometric quantitation), morphological (TEM, nm) and structural (protein NMR, spectra) characteristics useful to discriminate PD, DLB and MSA or different phenotypes of the same disease. It is known that there is a clinical and neuropathological heterogeneity among these diseases and this can be associated with the presence of different aberrant conformers of maS. Through in-depth analyses of the RT-QuIC reaction products we will evaluate whether these differences are useful to obtain patient stratification. .

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Moda, PHD, Principal Investigator — Fondazione IRCCS Istituto Neurologico Carlo Besta
Locations (3):
- Italy (3):
  - Consorzio Interuniversitario Risonanze Magnetiche Metallo Proteine (CIRMMP), Sesto Fiorentino, FI
  - IRCCS Centro San Giovanni di Dio, Brescia
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan

IPD SHARING:
Plan to Share IPD: Yes
e-CRF created with RedCap
Supporting Information: ICF